CLINICAL TRIAL: NCT05900635
Title: Effect of Adding Lactoferrin to Oral Iron Supplementation for the Treatment of Iron Deficiency Anemia in Chronic Kidney Disease Patients
Brief Title: Effect of Adding Lactoferrin on Oral Iron on Anemia in Chronic Kidney Disease Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107174
Record Dates: First submitted 2023-02-04; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-02

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: Lactoferrin; Anemia; Chronic Kidney Disease; Oral iron
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Lactoferrin; ferroglycine sulfate

STUDY DESIGN:
Intervention Model Description: Prospective, open-labeled, parallel, randomised controlled trial
Masking Description: open labeled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Patients in this group will initiate treatment with oral ferrous glycine sulfate (100mg) every other day for 3 months
  Interventions: Drug: Ferrous Glycine Sulfate
- Intervention (Active Comparator): Patients in this group will initiate treatment with oral lactoferrin (one sachet that contains 100mg) with oral ferrous glycine sulfate (100mg) every other day for 3 months
  Interventions: Drug: Lactoferrin; Drug: Ferrous Glycine Sulfate

INTERVENTIONS:
Drug: Lactoferrin — Effect of adding Lactoferrin to Oral Iron Supplementation for the treatment of Iron Deficiency Anemia in Chronic Kidney Disease Patients
  Arms: Intervention
Drug: Ferrous Glycine Sulfate — Effect of adding Lactoferrin to Oral Iron Supplementation for the treatment of Iron Deficiency Anemia in Chronic Kidney Disease Patients

SUMMARY:
The aim of this study is to evaluate the effects of adding lactoferrin to the every-other-day oral iron supplementation in iron deficiency anemia and chronic kidney disease patients.

DETAILED DESCRIPTION:
1. Ethical committee approval has been obtained from Ethics committee of Faculty of Medicine, Alexandria University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Sixty chronic kidney disease patients with iron defficiency anemia,will be recruited from the Kidney and Urology Center (KUC) and Alexandria main university hospital (AMUH).

   The 60 participants will be randomly assigned into 2 arms.

   Control arm (n=30): will be treated with oral ferrous glycine sulfate (100mg) every other day for 3 months

   Intervention arm (n=40): will be treated with oral lactoferrin (one sachet that contains 100mg) with oral ferrous glycine sulfate (100mg) every other day for 3 months.
4. All patients will be subjected directly at time of enrollment to the following; Complete history taking and demographic data (age, sex, …)
5. Blood samples will be drawn to measure the initial values of hemoglobin, hematocrit, serum iron, TIBC, Serum Transferrin Saturation (TSAT), and Hepcidin as primary outcome.
6. All patients will be followed up and treated during the study time. All relevant routine investigations and medications will be recorded.
7. At each visit, the subjects will be questioned about study compliance (diet and medications), concomitant medications, and adverse events.
8. The results obtained from the work will be tabulated and statistically analyzed using the appropriate statistical methods.
9. The findings will be discussed in view of the achievement of the aim, their significance and their comparison with other available works and information.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females aged ≥ 18 years old
2. Patients with eGFR ≥30 and ≤60 mL/min/1.73m2.
3. Absolute iron deficiency anemia (Hgb <10g/dL, serum ferritin <300ng/ml and Transferrin Saturation < 30% )

Exclusion Criteria:

1. Patients on intermittent hemodialysis (IHD)
2. Patients with any known cause of anemia other than iron deficiency or CKD (e.g., sickle cell anemia)
3. Patients who received EPO 4 weeks ago
4. Patients who received IV Iron 8 weeks ago
5. Patients who received blood Transfusion 8 weeks ago
6. Current history of GI bleeding
7. Malignancy history
8. Pregnancy or lactation in female participants
9. Patients non-adherent to at least 80% of the regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of the efficacy of the combination (lactoferrin plus ferrous glycine sulfate) versus ferrous glycine sulfate therapy in treatment of patients with iron deficiency anemia and CKD | 3 months
  Mean change in the level of Hemoglobin measured in gm/dl
Comparison of the efficacy of the combination (lactoferrin plus ferrous glycine sulfate) versus ferrous glycine sulfate therapy in treatment of patients with iron deficiency anemia and CKD | 3 months
  Mean change in the level of serum Iron measured in ug/mL
Comparison of the efficacy of the combination (lactoferrin plus ferrous glycine sulfate) versus ferrous glycine sulfate therapy in treatment of patients with iron deficiency anemia and CKD | 3 months
  Mean change in total iron binding capacity (TIBC) measured in ug/mL
Comparison of the efficacy of the combination (lactoferrin plus ferrous glycine sulfate) versus ferrous glycine sulfate therapy in treatment of patients with iron deficiency anemia and CKD | 3 months
  Mean change in serum transferrin saturation (TSAT) measured in %
Comparison of the efficacy of the combination (lactoferrin plus ferrous glycine sulfate) versus ferrous glycine sulfate therapy in treatment of patients with iron deficiency anemia and CKD | 3 months
  Mean change in serum hepcidin measured in ng/ml

SECONDARY OUTCOMES:
Evaluation of tolerability and gastrointestinal adverse events | 3 months
  The subjects will be contacted to be questioned about medications adherence and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F Elkoraie, Prof, Principal Investigator — Alexandria University; Magda A Elmassik, Prof, Principal Investigator — Alexandria University; Noha A Hamdy, PhD, Principal Investigator — Alexandria University; Engy M Emam, PharmD, Principal Investigator — Alexandria University
Locations (1):
- Kidney and Urology Center, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No